CLINICAL TRIAL: NCT02194556
Title: Sequential and Maintenance Icotinib Plus Chemotherapy Versus Icotinib Maintenance After Chemotherapy in Untreated Advanced Non-small-cell Lung Cancer: a Randomized, Open-label Study
Brief Title: Sequential and Maintenance Icotinib Plus Chemotherapy Versus Icotinib Maintenance After Chemotherapy in Advanced NSCLC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BD-IC-IV69
Record Dates: First submitted 2014-07-16; First posted 2014-07-18 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: EGFR Positive Non-small Cell Lung Cancer; Adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma | interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sequential and maintenance icotinib (Experimental): Patients are administered with sequential and maintenance icotinib plus chemotherapy. Gemcitabine 1000mg/m2 iv d1 and d8, cisplatin 75mg/m2 iv d1, icotinib 125 mg is administered orally three times per day at d 8-21, every 3 weeks for a cycle. After receiving a maximum of 4-cycle treatment, non-progressive patients continue to receive icotinib as maintenance treatment until disease progression or intolerable toxicity.
  Interventions: Drug: Sequential and maintenance icotinib
- Maintenance icotinib (Active Comparator): Gemcitabine 1000mg/m2 iv d1 and d8, cisplatin 75mg/m2 iv d1. After receiving a maximum of 4-cycle treatment, non-progressive patients continue to receive icotinib (125 mg three times per day) as maintenance treatment until disease progression or intolerable toxicity.
  Interventions: Drug: Maintenance icotinib

INTERVENTIONS:
Drug: Sequential and maintenance icotinib — Patients are administered with sequential and maintenance icotinib plus chemotherapy. Gemcitabine 1000mg/m2 iv d1 and d8, cisplatin 75mg/m2 iv d1, sequential icotinib 125 mg is administered orally three times per day at d 8-21, every 3 weeks for a cycle. After receiving a maximum of 4-cycle treatment, non-progressive patients continue to receive maintenance icotinib until disease progression or intolerable toxicity.
  Other Names: Gemzar; DDP; Comana, BPI-2009
  Arms: Sequential and maintenance icotinib
Drug: Maintenance icotinib — Gemcitabine 1000mg/m2 iv d1 and d8, cisplatin 75mg/m2 iv d1. After receiving a maximum of 4-cycle treatment, non-progressive patients continue to receive maintenance icotinib (125 mg three times per day) until disease progression or intolerable toxicity.
  Other Names: Gemzar; DDP; Comana, BPI-2009
  Arms: Maintenance icotinib

SUMMARY:
This randomised, controlled, open-label, prospective trial is designed to assess the efficacy and safety of icotinib maintenance therapy after sequential Icotinib plus chemotherapy versus Icotinib maintenance therapy after chemotherapy in stage IIIB/IV non-small cell lung cancer patients with EGFR mutation.

ELIGIBILITY:
Inclusion Criteria:

* Stage IV or IIIB advanced non-small cell lung cancer patients
* Positive EGFR Mutation
* Non-progressive disease after first-line gemcitabine/cisplatin therapy
* Measurable lesion according to RECIST 1.1 with at least one measurable lesion

Exclusion Criteria:

* Previous anti-EGFR (epidermal growth factor receptor) monoclonal antibody or small molecular agent such as gefitinib, erlotinib and so on
* Patients with wild-type EGFR
* Evidence of interstitial lung diseases
* Severe hypersensitivity to icotinib or any of the excipients of this product.
* Evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the subject to participate in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-07; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | 15 months
  A duration from randomization date to disease progression(as defined by RECIST) or death. If a participant are known to have progressed, the time to progression is defined as the time from the date of randomization to the date of progression. Otherwise, a participant will be censored at the last date they are known not to be progressed.

SECONDARY OUTCOMES:
Overall survival | 24 months
  Overall Survival is assessed via calculation of the time to death due to any cause. If a participant is known to have died, the time to death is defined as the time from the date of randomization to the date of death. Otherwise, a participant will be censored at the last date they are known to be alive.
Objective response rate | 24 months
  Number of subjects with confirmed objective response according to the Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
Adverse events | 24 months
  The number of patients who suffered adverse events, which is graded by NCI CTCAE version 4.0.
Disease control rate (DCR) | 24 months
  Disease control rate including complete response (CR) o，partial response (PR) , stable disease (SD)

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohua Hu, MD, Principal Investigator — First Affiliated Hospital of Guangxi Medical University
Locations (1):
- First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi, China